CLINICAL TRIAL: NCT03300648
Title: Treating Brain Swelling in Pediatric Cerebral Malaria
Acronym: TBS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Children's National Research Institute (Other); Nationwide Children's Hospital (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Maryland, Baltimore (Other); Kamuzu University of Health Sciences (Other)
Responsible Party: Principal Investigator, Terrie Taylor, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TBS; U01AI126610 (NIH)
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Malaria, Cerebral
Keywords: coma; pediatrics
MeSH Terms: conditions — Malaria, Cerebral; Coma | interventions — Respiration, Artificial; Saline Solution, Hypertonic

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three study arms.
Who Masked: Outcomes Assessor
Masking Description: Investigators assessing outcome will be blinded to the arm to which the participant was randomly assigned
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Usual care (No Intervention): Hospitalization in a high dependency pediatric unit with skilled nursing, intravenous artesunate followed by oral artemisinin combination therapy, intravenous fluids, nasogastric feeding, elevation of the head of the bed by 30 degrees
- Mechanical ventilation (Experimental): Hospitalization in a high dependency pediatric unit with skilled nursing, intravenous artesunate followed by oral artemisinin combination therapy, intravenous fluids, nasogastric feeding, elevation of the head of the bed by 30 degrees, along with intubation and mechanical ventilation for a maximum of 7 days
  Interventions: Other: Mechanical ventilation
- Hypertonic saline (Experimental): Hospitalization in a high dependency pediatric unit with skilled nursing, intravenous artesunate followed by oral artemisinin combination therapy, intravenous fluids, nasogastric feeding, elevation of the head of the bed by 30 degrees, along with intravenous 3% hypertonic saline for a maximum of 7 days
  Interventions: Drug: Hypertonic saline

INTERVENTIONS:
Other: Mechanical ventilation — Intubation and mechanical ventilation for a maximum of 7 days
  Arms: Mechanical ventilation
Drug: Hypertonic saline — Intravenous 3 percent hypertonic saline for a maximum of 7 days
  Arms: Hypertonic saline

SUMMARY:
This study evaluates the effectiveness of two interventions in Malawian children with cerebral malaria at high risk of death. One-third of the participants will receive treatment as usual, one-third will receive treatment as usual and be placed on a mechanical ventilator, and one-third will receive treatment as usual plus intravenous hypertonic saline.

DETAILED DESCRIPTION:
An important mechanism of death in children with cerebral malaria is diffuse cerebral swelling, cerebral herniation, compression of the brainstem respiratory center, and respiratory arrest. In those who survive their illness without specific interventions, reversal of diffuse cerebral swelling is rapid.

Mechanical ventilation may help to preserve life while diffuse brain swelling diminishes. Intravenous hypertonic saline may work as an osmotic diuretic, directly decreasing brain swelling.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral P. falciparum parasitemia of any density
* Blantyre Coma Score ≤2
* No evidence of meningitis on lumbar puncture
* Consciousness not regained after correction of hypoglycemia (if hypoglycemia is present)
* Male or female whose age on the day of screening is between 6 months and 12 years old
* Severely increased brain volume on magnetic resonance imaging
* Provision of consent by guardian
* Willingness to return for 1, 6, and 12 month post-randomization follow-up visits

Exclusion Criteria:

* Gross malnutrition as evidenced by peripheral edema, hair color changes, or severe wasting
* Advanced Human Immunodeficiency Virus (HIV) disease - defined as known HIV positive status and evidence of severe wasting
* Evidence of recent head trauma by history or physical examination
* Pneumonia as evidenced by oxygen saturation on room air of <85%
* Gastroenteritis and shock as evidenced by capillary refill >3 seconds or skin tenting

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terrie E Taylor, DO, Principal Investigator — Michigan State University
Locations (1):
- Queen Elizabeth Central Hospital, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data may be made available to other researchers
Time Frame: Starting 6 months after publication

REFERENCES:
- [Derived] Postels DG. Leveling the Playing Field: Combining Pediatric Neurology and Global Health. Pediatr Neurol. 2021 Jul;120:61-62. doi: 10.1016/j.pediatrneurol.2021.04.012. Epub 2021 Apr 25. No abstract available. PMID 34020114

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from 8 January 2018 through 24 May 2023. Children were recruited from Queen Elizabeth Central Hospital and were referred in from 6 surrounding District Hospitals, all in southern Malawi
Pre-assignment Details: Enrolled participants underwent screening brain magnetic resonance imaging. If the images showed highly increased brain volume (brain volume scores of 6-8) they were randomized to immediate ventilation, intravenous hypertonic saline, or treatment as usual (controls)
Groups:
- Mechanical Ventilation: Intubation and mechanical ventilation at the time of randomization
- Hypertonic Saline: Treatment as usual plus continuous infusion of intravenous 3 percent hypertonic saline
- Controls (Treatment as Usual): Treatment as usual
Period: Overall Study
Arm/Group | Mechanical Ventilation | Hypertonic Saline | Controls (Treatment as Usual)
Started | 23 | 17 | 17
Completed | 23 | 17 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mechanical Ventilation | Hypertonic Saline | Controls (Treatment as Usual) | Total
Number analyzed (Participants) | 23 | 17 | 17 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.1 (3.1) | 5.8 (4.1) | 6.5 (3.5) | 5.9 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 8 | 22
  Male | 15 | 11 | 9 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 23 | 17 | 17 | 57
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participant]
  Malawi | 23 | 17 | 17 | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Died
Description: Alive or dead
Time Frame: Within 7 days of randomization
Measure: Count of Participants; unit: Participants
Groups:
- Treatment as Usual: Treatment as usual
Arm/Group | Mechanical Ventilation | Hypertonic Saline | Treatment as Usual
Number analyzed (Participants) | 23 | 17 | 17
Participants | 5 | 5 | 5

2. Secondary Outcome: Neurodevelopmental Disability
Description: Presence and severity of neurodevelopmental disability in survivors
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Mechanical Ventilation | Hypertonic Saline | Controls (Treatment as Usual)
Number analyzed (Participants) | 18 | 12 | 12
Participants | 5 | 4 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Mechanical Ventilation | Hypertonic Saline | Controls (Treatment as Usual)
All-Cause Mortality (participants affected / at risk) | 5/23 | 5/17 | 5/17
Serious Adverse Events (participants affected / at risk) | 4/23 | 1/17 | 2/17
Other Adverse Events (participants affected / at risk) | 0/23 | 0/17 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mechanical Ventilation (N=23) | Hypertonic Saline (N=17) | Controls (Treatment as Usual) (N=17)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Respiratory problems from ventilator (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Low enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT03300648/Prot_SAP_000.pdf